CLINICAL TRIAL: NCT03293758
Title: Food and Microbiome Longitudinal Investigation (FAMiLI)
Status: Recruiting | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 12-00855; R21CA183887 (NIH)
Record Dates: First submitted 2017-09-22; First posted 2017-09-26 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Cancer; Cardiovascular Diseases
MeSH Terms: conditions — Neoplasms; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The NYU Human Microbiome Study Cohort is designed to improve understanding of the role of human microbiome in health and disease. This study will serve as a critical NYU biorepository resource for research on human genetics and the microbiome in health and disease

ELIGIBILITY:
Inclusion Criteria:

* Age > 40

Exclusion Criteria:

* Use of long term antibiotics.
* Pregnant

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects in the United States identified at NYU clinics, community organizations, and online participant databases.
Sampling Method: Non-Probability Sample
Enrollment: 14000 (Estimated)
Dates: Start 2016-05-16 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Demographic | 5 Years
  sex, race, education, oral health status, lifestyle, medical history, anthropometry, and medication use will be collected using the baseline questionnaire at enrolment. The collected information will provide risk stratification information for statistical control in studies of colorectal tumors and other major chronic diseases.

SECONDARY OUTCOMES:
Differences in human microbiota between subjects with colorectal adenoma or colorectal cancer and those without. | 5 Years
  Pairwise alignment and clustering of sequences into operational taxonomic units (OTUs)

CONTACTS AND LOCATIONS:
Overall Officials: Jiyoung Ahn, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States